CLINICAL TRIAL: NCT04203641
Title: A Phase Ib/II Study of the Microenvironment Modifier L-DOS47 Plus Doxorubicin for the Treatment of Patients With Previously Treated Advanced Pancreatic Cancer
Brief Title: L-DOS47 Plus Doxorubicin in Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The primary reason for early termination was budget constraint.
Sponsor: Helix BioPharma Corporation (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LDOS006
Record Dates: First submitted 2019-09-16; First posted 2019-12-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-10

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; immunoconjugate; tumor microenvironment alkalinization
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm study that includes an initial three cohort dose escalation phase with 3, 6 and 9 µg/kg of L-DOS47 in combination with doxorubicin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-DOS47 + doxorubicin (Experimental): Patients will be recruited into escalating dosing cohorts of 3, 6 and 9 µg/kg of L-DOS47, with a minimum of 3 and a maximum of 6 patients per cohort. A fixed dose of intravenous doxorubicin [20 mg/m2/week] will be administered in combination with L-DOS47 across all cohorts.
  Interventions: Biological: L-DOS47; Drug: Doxorubicin

INTERVENTIONS:
Biological: L-DOS47 — A treatment cycle will be 28 days, with patients receiving L-DOS47 on Days 1, 8, 15, and 22.
Drug: Doxorubicin — A treatment cycle will be 28 days, with patients receiving doxorubicin on Days 2, 9, 16 and 23

SUMMARY:
This study will evaluate the safety and tolerability of escalating doses of L-DOS47 in combination with doxorubicin, as well as preliminary anti-tumor activity in patients with previously treated advanced pancreatic cancer.

DETAILED DESCRIPTION:
The Phase Ib part of the study will apply a standard 3 + 3 algorithm for dose escalation to determine the appropriate L-DOS47 maximum tolerated dose to use in combination with doxorubicin for the Phase II part of the study. Patients will be recruited into 3 cohorts where each cohort will receive increasing weekly dose levels of L-DOS47 in combination with a fixed dose of 20 mg/m2 of doxorubicin weekly. The decision for escalation to the next dose level will be made after all patients in a cohort have completed 4 weeks of combination treatment and the safety data have been reviewed by the Safety Review Committee. If a patient in any cohort experiences a dose limiting toxicity, an additional 3 patients will be enrolled, for a maximum of up to 18 patients in this initial dose escalation part of the study.

The Phase II part of the study will focus on evaluating preliminary anti-tumor activity, as well as continuing to evaluate safety and tolerability of L-DOS47 in combination with doxorubicin. A further 11 additional patients will be enrolled in this phase of the study, which is designed to ensure patient safety and to detect whether there is a level of anti-tumor activity that would be worth pursuing in a larger clinical trial. Patients will be initiated on the L-DOS47 dose determined in Phase I, in combination with 20 mg/m2 doxorubicin, with tumor marker carbohydrate antigen 19-9 (CA19-9) measurements at each treatment cycle, and radiological assessments every two treatment cycles.

Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

Safety will be assessed by reported adverse events (AEs), serious adverse events (SAEs), physical exams, vital signs, Karnofsky Performance Status, electrocardiogram (ECG), echocardiogram (ECHO)/multigated acquisition scan (MUGA), clinical laboratory evaluations (hematology, chemistry, coagulation and urinalysis), and anti-L-DOS47 antibody levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years old
2. One or more metastatic tumors measurable on computed tomography (CT) scan per RECIST version 1.1 and screening FDG-PET scan with maximum standardized uptake value (SUV max) ≥ 5.5 for at least one lesion consistent with pancreatic cancer.
3. Karnofsky performance status ≥ 70%
4. Life expectancy of at least 3 months
5. Able to understand the information provided to them and to give written institutional review board (IRB)-approved informed consent prior to any study activities being conducted
6. A negative pregnancy test (if of child bearing potential)
7. Acceptable liver function:

   1. Bilirubin ≤ 1.5 times upper limit of normal
   2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and Alkaline phosphatase (ALP) ≤ 2.5 times upper limit of normal (ULN; if liver metastases are present, then ≤ 5 x ULN is allowed)
8. Acceptable renal function as defined by creatinine ≤1.5x institutional upper limits of normal, or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
9. Acceptable hematologic status:

   1. Granulocyte ≥ 1500 cells/mm3
   2. Platelet count ≥ 100,000 (plt/mm3)
   3. Hemoglobin ≥ 9g/dL
10. Urinalysis:

    a) No clinically significant abnormalities
11. Acceptable coagulation status

    1. Prothrombin time within 1.5x of normal limits
    2. Partial thromboplastin time (PTT) within 1.5x of normal limits
12. For men and women of child-bearing potential, the use of effective contraceptive methods during the study
13. Normal ejection fraction on ECHO or MUGA

Exclusion Criteria:

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
2. Abnormal ejection fraction on ECHO or MUGA
3. Active, uncontrolled bacterial, viral, or fungal infections requiring systematic therapy
4. Pregnant or nursing women. NOTE: Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
5. Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 3 weeks prior to study entry
6. Major surgery within 4 weeks prior to study entry
7. Unwillingness or inability to comply with procedures required in this protocol
8. Known infection with HIV, hepatitis B, or hepatitis C
9. Serious nonmalignant disease (eg hydro nephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
10. Patients who are currently receiving any other investigational agent
11. Patients with any evidence of uncontrolled brain metastases or carcinomatosis meningitis.
12. Patients with marked screening prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval > 480 milliseconds (CTCAE grade 1) using Fredericia's QT correction formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Number of complete plus partial responders as per RECIST version 1.1 | 24 weeks
  Assess number of complete plus partial responders according to RECIST version 1.1 as a measure of preliminary anti-tumor activity of L-DOS47 in combination with doxorubicin
Adverse events (as per CTCAE v. 5.0) | 24 weeks
  Assess frequency of treatment emergent adverse events as per Common Terminology Criteria for Adverse Events (CTCAE) v. 5 as a measure of safety and tolerability of L-DOS47 in combination with doxorubicin

SECONDARY OUTCOMES:
Change in tumor pH | From screening to end of Cycle 2, where each treatment cycle is 28 days.
  Change from screening tumor pH as measured by SUV on fluorodeoxyglucose-positron emission tomography scan (FDG-PET) scan
Carbohydrate antigen (CA) 19-9 biomarker level | Up to 24 weeks
  Change from screening in CA19-9 biomarker levels
Proportion of patients expressing anti-L-DOS47 antibodies | Up to 24 weeks
  Assess number of patients expressing anti-L-DOS47 antibodies levels as a measure of

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — Scottsdale Healthcare Hospitals DBA HonorHealth
Locations (3):
- United States (3):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - Atlantic Health System, Morristown Medical Center, Morristown, New Jersey
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin